CLINICAL TRIAL: NCT01522079
Title: Spinal Muscular Atrophy and Cardiac Autonomic Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Principal Investigator, Cristina Marcia Dias, Professor DSc, Centro Universitário Augusto Motta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dias
Record Dates: First submitted 2012-01-24; First posted 2012-01-31 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Spinal Muscular Atrophy
Keywords: spinal muscular atrophy; heart rate variability; posture; air stacking
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Air stacking (Experimental): Electrocardiogram signals were recorded for analyses of heart rate variability during air stacking in supine and sitting position.
  Interventions: Procedure: Air stacking manuever

INTERVENTIONS:
Procedure: Air stacking manuever — Electrocardiogram signals were recorded for analyses of heart rate variability during air stacking in supine and sitting position
  Other Names: HRV during air stacking

SUMMARY:
Respiratory dysfunction is the major cause of morbidity and mortality in patients with spinal muscular atrophy (SMA). Air stacking is a clearance airway technique frequently used but its effects on cardiac autonomic function in patients with spinal muscle atrophy is not clear.

Objective: To evaluate the acute effect of air stacking and posture on cardiac autonomic function in patients with spinal muscular atrophy types II and III.

Methods: Patients with spinal muscle atrophy type II and III will be recruited. Electrocardiogram signals will be recorded for analyses of heart rate variability during air stacking in supine and sitting position.

DETAILED DESCRIPTION:
Background: Respiratory dysfunction is the major cause of morbidity and mortality in patients with spinal muscular atrophy. Air stacking is a clearance airway technique frequently used but its effects on cardiac autonomic function in patients with spinal muscle atrophy is not clear.

Objective: To evaluate the acute effect of air stacking and posture on cardiac autonomic function in patients with spinal muscular atrophy types II and III.

Methods: Patients with spinal muscle atrophy type II and III will be recruited. Electrocardiogram signals will be recorded for analyses of heart rate variability during air stacking in supine and sitting position. Data will collected before, during and after air stacking and will be compared using Anova Repeated Measures or Kruskal-Wallis Anova on Ranks, followed by Tukey test. The relationship between heart rate variability indexes and age will be evaluated by Pearson correlation. Significant level will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SMA types II and III,
* absence of acute respiratory disease in the last two weeks,
* agreement to participate in the study,
* according written informed consent and
* at least 5 years old.

Exclusion Criteria:

* respiratory disease in the last two weeks

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Cardiac autonomic function | Thirty minutes during air stacking manuever
  Evaluation of heart rate variability in patients with spinal muscular atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Cristina M Dias, PT - PhD, Principal Investigator — Centro Universitário Augusto Motta